CLINICAL TRIAL: NCT05625945
Title: Physical Activity Levels and Statin Therapy: Differences Between Symptomatic and Asymptomatic Statin Users
Brief Title: Physical Activity Levels and Statin Therapy
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL9196
Record Dates: First submitted 2022-10-23; First posted 2022-11-23 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Cardiovascular Diseases; HMG COA Reductase Inhibitor Adverse Reaction; Muscle Pain
MeSH Terms: conditions — Cardiovascular Diseases; Myalgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Symptomatic statin users: Statin users with self-reported muscle symptoms
  Interventions: Behavioral: Physical activity monitoring
- Asymptomatic statin users: Statin users without muscle symptoms
  Interventions: Behavioral: Physical activity monitoring

INTERVENTIONS:
Behavioral: Physical activity monitoring — Physical activity patterns will be measured using the activPAL3 micro monitor

SUMMARY:
Rationale: Combining statin treatment and physical activity is very effective for the prevention of cardiovascular diseases. Statins are well-tolerated by most patients, but may cause statin-associated muscle symptoms (SAMS).

Objective: To identify predictors for SAMS in statin users and to objectively assess physical activity levels and sedentary time between symptomatic and asymptomatic statin users.

DETAILED DESCRIPTION:
Combining statin treatment and physical activity is very effective for the prevention of cardiovascular diseases. Statins are well-tolerated by most patients, but may cause statin-associated muscle symptoms (SAMS). Physical activity may exacerbate SAMS, producing decreased physical activity levels or statin nonadherence. However, it is unknown if daily activity patterns differ between symptomatic and asymptomatic statin users.

In this cross-sectional observational study the investigators will assess if physical activity levels and sedentary time differ between symptomatic and asymptomatic statins users. Secondly, questionnaires will be used to assess predictors of SAMS.

ELIGIBILITY:
Inclusion Criteria:

* Mentally able to give informed consent
* Statin treatment for at least 3 months

Exclusion Criteria:

* Known hereditary muscle defect
* Known mitochondrial disease
* Other diseases known to cause muscle symptoms (e.g. m. Parkinson or rheumatic diseases)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic statin users (n=100) and asymptomatic statin users (n=100)
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2023-11-16 (Actual)

PRIMARY OUTCOMES:
Physical activity | during 1 week
  Physical activity (min/day) will be assessed using the activPAL3 micro monitor
Sedentary time | during 1 week
  Sedentary time (min/day) will be assessed using the activPAL3 micro monitor

SECONDARY OUTCOMES:
Predictors of statin-associated muscle complaints (SAMS) | 1 moment (cross-sectional)
  Using questionnaires predictors of SAMS will be explored

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physiology, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No